CLINICAL TRIAL: NCT04669145
Title: Single-Shot Versus Continuous Regional Anesthesia for Treating Acute Postoperative Pain in Pediatric Orthopaedic Surgery: A Prospective Randomized Trial
Brief Title: Regional Anesthesia in Pediatric Orthopaedic Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.403
Record Dates: First submitted 2020-12-06; First posted 2020-12-16 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia, Local; Anesthesia; Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Continuous Regional Anesthesia Lower Limb Surgery (Experimental): Various types of regional anesthesia blocks will be performed based on the patient's injuries including fascia iliaca plane blocks, femoral nerve blocks, adductor canal blocks, popliteal approach sciatic nerve blocks, and saphenous nerve blocks A catheter will be placed for the given block for 48 hours. Those patients undergoing lower limb orthopaedic surgery will be randomized into single shot or continuous (catheter) regional anesthesia.
  Interventions: Drug: Ropivacaine
- Single Shot Regional Anesthesia Lower Limb Surgery (Experimental): Various types of regional anesthesia blocks will be performed based on the patient's injuries including fascia iliaca plane blocks, femoral nerve blocks, adductor canal blocks, popliteal approach sciatic nerve blocks, and saphenous nerve blocks. These blocks will be given via a single dose or "single shot". Those patients undergoing lower limb orthopaedic surgery will be randomized into single shot or continuous (catheter) regional anesthesia.
  Interventions: Drug: Ropivacaine
- Continuous Regional Anesthesia Upper Limb Surgery (Experimental): Various types of regional anesthesia blocks involving the brachial plexus will be performed based on the patient's injuries. A catheter will be placed for the given block for 48 hours. Those patients undergoing upper limb orthopaedic surgery will be randomized into single shot or continuous (catheter) regional anesthesia.
  Interventions: Drug: Ropivacaine
- Single Shot Regional Anesthesia Upper Limb Surgery (Experimental): Various types of regional anesthesia blocks involving the brachial plexus will be performed based on the patient's injuries. A catheter will be placed for the given block for 48 hours. Those patients undergoing upper limb orthopaedic surgery will be randomized into single shot or continuous (catheter) regional anesthesia.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Dosing and volume will vary based on type of block used and weight of patient because of the pediatric population in the study.

SUMMARY:
To identify the benefits from regional anesthesia use as pain management in the pediatric population by delineating the differences in efficacy of continuous nerve blockade versus single-shot techniques after pediatric orthopaedic limb procedures. By doing this, the investigators can determine if specific anesthetic techniques should become a standard of care in pain management for the pediatric population and supersede the need for opioid medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary orthopaedic limb surgery
* Outpatient orthopaedic surgeries
* Patients undergoing orthopaedic surgery who would normally receive regional anesthesia

Exclusion Criteria:

* Patients younger than 5 years of ago or older than 18 years of age
* Revision orthopaedic surgeries
* Spinal orthopaedic surgeries
* Orthopaedic surgeries where the standard of care for type of regional anesthesia has been established (continuous regional for ACL reconstruction)
* Patients with the inability to articulate pain scores
* Inpatient orthopaedic surgeries
* Patients undergoing orthopaedic limb surgery with risk of compartment syndrome (i.e. acute supracondylar humerus fractures)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | For first 48 hours post-operatively.
  Amount of opioid medications taken for pain control.

SECONDARY OUTCOMES:
Opioid Consumption | Through 12 hours post-operatively.
  Amount of opioid medications taken for pain control.
Opioid Consumption | Through 24 hours post-operatively.
  Amount of opioid medications taken for pain control.
Opioid Consumption | Through 36 hours post-operatively.
  Amount of opioid medications taken for pain control.
Opioid Consumption | Through 48 hours week post-operatively.
  Amount of opioid medications taken for pain control.
Opioid Consumption | Through 72 hours post-operatively.
  Amount of opioid medications taken for pain control.
Opioid Consumption | Through 96 hours post-operatively.
  Amount of opioid medications taken for pain control.
Opioid Consumption | Through 120 hours post-operatively.
  Amount of opioid medications taken for pain control.
Opioid Consumption | Through 144 hours post-operatively.
  Amount of opioid medications taken for pain control.
Opioid Consumption | Through 168 hours post-operatively.
  Amount of opioid medications taken for pain control.
Emergency Room Visits | Within 2 weeks post-operatively.
  Emergency room visits due to poor pain control.
Pain Scores | At 12 hours post-operatively.
  Universal Pain Assessment tool will be used. The pain scale ranges from 0 to 10 with 0 being no pain and 10 being the worst possible pain.
Pain Scores | At 24 hours post-operatively.
  Universal Pain Assessment tool will be used. The pain scale ranges from 0 to 10 with 0 being no pain and 10 being the worst possible pain.
Pain Scores | At 36 hours post-operatively.
  Universal Pain Assessment tool will be used. The pain scale ranges from 0 to 10 with 0 being no pain and 10 being the worst possible pain.
Pain Scores | At 48 hours post-operatively.
  Universal Pain Assessment tool will be used. The pain scale ranges from 0 to 10 with 0 being no pain and 10 being the worst possible pain.
Pain Scores | At 72 hours post-operatively.
  Universal Pain Assessment tool will be used.The pain scale ranges from 0 to 10 with 0 being no pain and 10 being the worst possible pain.
Pain Scores | At 96 hours post-operatively.
  Universal Pain Assessment tool will be used.The pain scale ranges from 0 to 10 with 0 being no pain and 10 being the worst possible pain.
Pain Scores | At 120 hours post-operatively.
  Universal Pain Assessment tool will be used.The pain scale ranges from 0 to 10 with 0 being no pain and 10 being the worst possible pain.
Pain Scores | At 144 hours post-operatively.
  Universal Pain Assessment tool will be used.The pain scale ranges from 0 to 10 with 0 being no pain and 10 being the worst possible pain.
Pain Scores | At 168 hours post-operatively.
  Universal Pain Assessment tool will be used.The pain scale ranges from 0 to 10 with 0 being no pain and 10 being the worst possible pain.
Pain Scores | At 2 weeks post-operatively.
  Universal Pain Assessment tool will be used. The pain scale ranges from 0 to 10 with 0 being no pain and 10 being the worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Medical Center, Jefferson, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No